CLINICAL TRIAL: NCT02701205
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Safety and Efficacy Study of Recombinant Human TNF Receptor-IgG Fusion Protein for Injection (Qiangke®) to Treat Moderate to Severe Plaque Psoriasis
Brief Title: Safety and Efficacy Study of Etanercept (Qiangke®) to Treat Moderate to Severe Plaque Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Celgen Bio-Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QRSTPP
Record Dates: First submitted 2016-02-28; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Plaque Psoriasis; Psoriasis
Keywords: Plaque Psoriasis; Skin Disease
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- etanercept (Experimental): Recombinant Human TNF Receptor-Ig Fusion Protein for Injection（Qiangke®) 50mg twice a week for 12 weeks, then Two vials of Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 25mg twice a week from Week 12 to Week 24
  Interventions: Biological: etanercept
- etanercept (half dose) (Experimental): One vial of Recombinant Human TNF Receptor-Ig Fusion Protein for Injection（Qiangke®） 25mg and one vial of placebo twice a week for 12 weeks, then Two vials of Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 25mg twice a week from Week 12 to Week 24
  Interventions: Biological: etanercept (half dose)
- Placebo (Placebo Comparator): Two vials of Placebo twice a week for 12 weeks, then Two vials of Recombinant Human TNF Receptor-Ig Fusion Protein for Injection（Qiangke®) 25mg twice a week from Week 12 to Week 24
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: etanercept — Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 50mg twice a week by subcutaneous injection for 12 weeks, At the end of the first 12 weeks, all subjects will be treated with Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 50 mg once a week for an additional 12 weeks.
  Other Names: Qiangke®
  Arms: etanercept
Biological: etanercept (half dose) — Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 25mg twice a week by subcutaneous injection for 12 weeks, At the end of the first 12 weeks, all subjects will be treated with Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 50 mg once a week for an additional 12 weeks.
  Other Names: Qiangke®
  Arms: etanercept (half dose)
Drug: placebo — two vials of placebo twice a week by subcutaneous injection for 12 weeks, At the end of the first 12 weeks, all subjects will be treated with Recombinant Human TNF Receptor-Ig Fusion Protein for Injection 50 mg once a week for an additional 12 weeks.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multicentral clinical trial to investigate the efficacy and safety of Recombinant Human TNF Receptor-Ig Fusion Protein for Injection (Qiangke®) in the treatment of Moderate to Severe Plaque Psoriasis. The primary purpose is to assess the different maintaining treatment programme in Moderate to Severe plaque psoriasis by Qiangke®. And the second purpose is to assess the efficacy and safety of Qiangke® in Moderate to Severe Plaque Psoriasis. The trial will include 216 Moderate to Severe plaque psoriasis patients,and at the first stage they will be randomized divided into three group: full-dose of Qiangke® group, half-dose of Qiangke® group and placebo group.And the blind stage will last for 12 weeks. Then at the second stage, all patients will receive 50mg qw of Qiangke® for additional 12 weeks.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease that can lead to significant physical and psychologic distress for patients.Recombinant Human TNF Receptor-Ig Fusion Protein for Injection (Qiangke®) can block the role of the cytokine tumor necrosis factor (TNF)-alpha.

TNF-α plays a major role in the pathophysiology of both Psoriasis（PsO）and Psoriatic Arthritis (PsA). TNF-α levels are elevated in psoriatic skin lesions, serum samples, and synovial fluid. Anti-TNF-α therapy has shown efficacy in treating psoriatic skin lesions, joint pain and swelling, enthesitis, and dactylitis plus the ability to improve mobility, reduce radiographic progression of disease, and influence quality of life parameters.

Qiangke® is a dimeric, soluble fusion protein consisting of the extracellular ligand binding portion of the TNF receptor linked to the Fc portion of human Immunoglobulin gamma-1（IgG1）. It is capable of binding and neutralizing soluble TNF and transmembrane TNF. It alters neutrophil migration and dendritic cell and T-cell maturation and migration, thus decreasing the local and systemic production of pro-inflammatory cytokines and their subsequent effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, age 18-65,Asian.
2. Freely provides both verbal and written informed consent.
3. Consent to use effective contraception during the trial period.
4. Participant had a clinical diagnosis of psoriasis for at least 6 months, and had moderate to severe plaque psoriasis
5. Participant must have a Psoriasis Area Severity Index score greater than or equal to 12 at the baseline visit and Body Surface Area involvement greater than or equal to 10% at the baseline visit.
6. Participant has previous exposure to systemic psoriasis therapy or phototherapy, but not ideal.
7. Meet the following criteria for Tuberculosis screening: A. has no prior history of occult or active tuberculosis. B. No signs or symptoms of active tuberculosis in history and / or physical examination. C. in the first 6 weeks of the trial, tuberculosis screening test meet the requirements of the trial.
8. Laboratory screening results:Hemoglobin≥110g/L.White blood cell≥4 * 109 /L. Neutrophil≥1.5 * 109/L.Platelet≥100 * 109/L.Serum alanine aminotransferase and / or aspartate aminotransferase not more than 1.5 times of the upper limit of normal.Serum creatinine does not exceed 1.5 mg/dL (International units: ≤133 mol/L).
9. During the first 2 weeks of the study, Participant must stop adjuvant therapy including traditional Chinese medicine and acupuncture.
10. Hepatitis B (HBV) screening in compliance with the requirements of this test.
11. Weight≥60Kg.

Exclusion Criteria:

1. Pustular, erythrodermic, and/or guttate forms of psoriasis.
2. Participant had treated with TNF antagonists within 6 weeks prior to the Baseline visit.
3. Participant had treated with Other biological agents within 6 weeks prior to the Baseline visit.
4. Participant had treated with Phototherapy or systemic antipsoriatic treatment (such as:Methotrexate（MTX）， acitretin, cyclosporine, Total Glucosides of Paeony（TGP）, treatment of psoriasis related Chinese medicines, etc.) and systemic corticosteroid treatment within 4 weeks prior to the Baseline visit.
5. Participant had treated with Topical corticosteroid therapy, vitamin A or D analogue or Anthralin within 2 weeks prior to the Baseline visit.
6. Participant received any drug that the drug's metabolism was less than 7 half lives before the Baseline visit.
7. Participant plans to pregnant or breast feeding or father during the study.
8. The history of occult or active granuloma infections, including histoplasmosis, coccidioidomycosis.
9. Participant has suffered from Non Mycobacterium tuberculosis infection or opportunistic infections (such as cytomegalovirus sense of dyeing, Pneumocystis carinii pneumonia, aspergillosis) within 6 weeks prior to the Baseline visit.
10. The close contact history of active tuberculosis patients or Tuberculosis screening results do not meet the requirements.
11. Participant has suffered from severe infection (for example hepatitis, pneumonia, acute pyelonephritis or sepsis), or participant use intravenous antibiotics now because of infection within 6 weeks prior to the Baseline visit.
12. Participant has suffered from chronic or recurrent infections before or at present, including (but not limited to) chronic kidney infection disease and chronic chest infectious diseases (such as bronchial dilation), sinusitis, recurrent urinary tract infections (such as recurrent pyelonephritis and chronic non remission cystitis), open, overflow liquid or infection of skin wound or ulcer.
13. Human immunodeficiency virus (HIV) antibody positive.
14. Hepatitis B virus (HBV) screening results do not meet the requirements.
15. Hepatitis C virus (HCV) antibody positive.
16. Participant has demyelinating diseases such as multiple sclerosis or optic neuritis.
17. A history of congestive heart failure, including asymptomatic congestive heart failure.
18. A history or sign of a lymph node hyperplasia, including lymphoma or suggestive of a possible sign such as the size and location of an enlarged lymph node or a history of clinically significant enlargement of the spleen.
19. Participant has symptoms or signs of severe, progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, nerve, mental or brain diseases.
20. There is a history of malignancy or previous history.
21. Joint prosthesis has not yet been removed or replaced.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 75% Reduction (PASI 75) Response at Week 12 | Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI 90 & 50 | Week 12
Proportion of subjects achieving PASI 90 & 50 & 75 | Week 24
Physician's Global Assessment (PGA) | Week 12 & 24
Nail Psoriasis Severity Index (NAPSI) | Week 12 & 24
Dermatology Life Quality Index (DLQI) | Week 12 & 24
Patient's Global Assessment (PGA) | Week 12 & 24

OTHER OUTCOMES:
Safety parameters - Number of Participants With Abnormal Laboratory Values and/or Adverse Events | Week 12 & 24
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhong Jin, M.D., Principal Investigator — Chinese Academy of Medical Sciences Peking Union Medical College
Locations (4):
- China (4):
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Institute of Dermatology and Skin Disease Hospital Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Changhai Hospital of The Second Military Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gottlieb AB, Chamian F, Masud S, Cardinale I, Abello MV, Lowes MA, Chen F, Magliocco M, Krueger JG. TNF inhibition rapidly down-regulates multiple proinflammatory pathways in psoriasis plaques. J Immunol. 2005 Aug 15;175(4):2721-9. doi: 10.4049/jimmunol.175.4.2721. PMID 16081850
- [Background] Gudjonsson JE, Elder JT. Psoriasis: epidemiology. Clin Dermatol. 2007 Nov-Dec;25(6):535-46. doi: 10.1016/j.clindermatol.2007.08.007. PMID 18021890
- [Background] Gupta MA, Gupta AK. Depression and suicidal ideation in dermatology patients with acne, alopecia areata, atopic dermatitis and psoriasis. Br J Dermatol. 1998 Nov;139(5):846-50. doi: 10.1046/j.1365-2133.1998.02511.x. PMID 9892952
- [Result] Leonardi CL, Powers JL, Matheson RT, Goffe BS, Zitnik R, Wang A, Gottlieb AB; Etanercept Psoriasis Study Group. Etanercept as monotherapy in patients with psoriasis. N Engl J Med. 2003 Nov 20;349(21):2014-22. doi: 10.1056/NEJMoa030409. PMID 14627786
- [Result] Kivelevitch D, Mansouri B, Menter A. Long term efficacy and safety of etanercept in the treatment of psoriasis and psoriatic arthritis. Biologics. 2014 Apr 17;8:169-82. doi: 10.2147/BTT.S41481. eCollection 2014. PMID 24790410
- [Result] Papp KA, Tyring S, Lahfa M, Prinz J, Griffiths CE, Nakanishi AM, Zitnik R, van de Kerkhof PC, Melvin L; Etanercept Psoriasis Study Group. A global phase III randomized controlled trial of etanercept in psoriasis: safety, efficacy, and effect of dose reduction. Br J Dermatol. 2005 Jun;152(6):1304-12. doi: 10.1111/j.1365-2133.2005.06688.x. PMID 15948997
- [Result] Sterry W, Ortonne JP, Kirkham B, Brocq O, Robertson D, Pedersen RD, Estojak J, Molta CT, Freundlich B. Comparison of two etanercept regimens for treatment of psoriasis and psoriatic arthritis: PRESTA randomised double blind multicentre trial. BMJ. 2010 Feb 2;340:c147. doi: 10.1136/bmj.c147. PMID 20124563
- [Result] Chiu HY, Wang TS, Cho YT, Tsai TF. Etanercept use for psoriasis in Taiwan: a case series study. Int J Dermatol. 2013 Jun;52(6):673-80. doi: 10.1111/j.1365-4632.2011.05273.x. Epub 2012 Feb 20. PMID 22348620